CLINICAL TRIAL: NCT01946737
Title: Diagnostic Performance of 64 Slice High Definition Computed Tomographic Coronary Angiography in Patients With High Risk of Significant Coronary Artery Disease.
Brief Title: High Definition CT Coronary Angiography Accuracy Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Plymouth NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Diagnostic
Other Study IDs: 11/P/050; 11/H0206/5 (Other: UK REC Reference Number)
Record Dates: First submitted 2013-09-03; First posted 2013-09-20 (Estimated); Last update posted 2013-09-20 (Estimated); Status verified 2013-09

CONDITIONS: Coronary Artery Disease
Keywords: Coronary; Artery; Disease; Diagnostic; Performance; Angiography
MeSH Terms: conditions — Coronary Artery Disease; Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Invasive coronary angiography (ICA) (Active Comparator): Routine diagnostic ICA
  Interventions: Radiation: Active Comparator: Invasive coronary angiography (ICA)
- HD-CTCA with ASIR (Experimental): HD-CTCA with Adaptive statistical iterative reconstruction (ASIR)within 4 weeks of routine diagnostic ICA
  Interventions: Radiation: HD-CTCA with Adaptive statistical iterative reconstruction (ASIR)

INTERVENTIONS:
Radiation: HD-CTCA with Adaptive statistical iterative reconstruction (ASIR)
  Arms: HD-CTCA with ASIR
Radiation: Active Comparator: Invasive coronary angiography (ICA)
  Arms: Invasive coronary angiography (ICA)

SUMMARY:
CT technology is evolving at a rapid pace, with introduction of multidetector row CT scanners (MDCT) and electrocardiographic (ECG) gating resulting in increasing numbers of heart scans CTCA (CT Coronary Angiography). CTCA provides a noninvasive alternative to conventional invasive coronary angiography (ICA), which is considered the gold standard in the investigation of coronary disease. There has been a gradual increase in the utilization of CTCA for primary assessment of low and intermediate risk patients. However concerns regarding radiation exposure and diagnostic accuracy, especially in the highrisk group, have prevented its widespread dissemination.

To achieve best possible temporal resolution (minimize cardiac motion artifacts) and spatial resolution (provide diagnostic accuracy) relatively high radiation exposure is required, as a result of its inverse relationship with image noise and resolution. However radiation (X-ray) is associated with increased risk of cancer in exposed patients and it is therefore essential to continually devise strategies to reduce radiation exposure whilst maintaining image quality.

A state-of-art CT scanner (Discovery CT750 HD, General Electric (GE) Healthcare), has been installed at Derriford hospital for further research on CTCA. It uses novel method of scanning, High Definition Computed Tomographic Coronary Angiography(HD-CTCA), analogous to high definition television) and image reconstruction (Adaptive Statistical Iterative Reconstruction ASIR)as opposed to conventional CT scanners using Filtered Back Projection (FBP)reconstruction. HD-CTCA enables acquisition of sharper images and ASIR offsets the resultant increase in radiation exposure. This is likely to result in images of higher diagnostic quality with an equivalent or slightly lower radiation exposure compared to present technology. Although initial results are encouraging, this needs further assessment before being applied to routine clinical practice. To assess this we have designed a study to perform HD-CTCA on 300 consecutive patients undergoing diagnostic ICA at Derriford hospital, directly comparing the accuracy of HD-CTCA to ICA (presently considered the gold standard).

Hypotheses:

There is no significant difference in the sensitivity and specificity of HD-CTCA for the detection of coronary artery stenosis of 50% or greater compared to conventional ICA.

ELIGIBILITY:
Inclusion Criteria:

* Patients > 40 years of age.
* Suspected or known coronary artery disease
* Admitted for diagnostic ICA

Exclusion Criteria:

* Consent cannot be obtained
* Age <40 years
* New York Heart Association (NYHA) Functional Classification - class III or IV heart failure
* Emergency imaging required (not enough time to consider the trial)
* Allergy to iodinated contrast or previous contrast induced nephropathy
* Intolerance to betablockers
* Uncontrolled rhythm disturbances (not suitable for CTCA)
* Serum Creatinine >200 micro mol/L within two weeks prior to procedure or chronic renal failure on dialysis

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 302 (Actual)
Dates: Start 2011-04; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Diagnostic accuracy of HD-CTCA for the detection of at least moderate stenosis (>50%) as defined on invasive coronary angiography in the high-risk target population. | 4 weeks
  We designed the New Generation Computed Tomographic Coronary Angiography (NG-CTCA) study to assess the diagnostic accuracy of high-definition CT with iterative reconstruction in an unselected population of patients suitable for CTCA with either a high pre-test probability of, or established coronary artery disease. Our hypothesis is that NGCT has a comparable diagnostic performance to invasive coronary angiography (ICA), using this as the reference standard

SECONDARY OUTCOMES:
The diagnostic accuracy of HD-CTCA for the detection of severe stenosis (70%) as defined by invasive coronary angiography. | 4 weeks

OTHER OUTCOMES:
The radiation dose delivered by HD-CTCA | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Carl Roobottom, BSc, MBChB(hon), MRCP. FRCR, Study Chair — University Hospital Plymouth NHS Trust; Srikanth Iyengar, MBBS, MS, FRCS, FRCR, Principal Investigator — University Hospital Plymouth NHS Trust
Locations (1):
- Plymouth Hospitals NHS Trust, Plymouth, Devon, United Kingdom